CLINICAL TRIAL: NCT05681923
Title: Platform for the Prospective Mother-child Study of the Determinants of Autism Spectrum Disorder and Neurodevelopmental Disorders Neurodevelopmental Disorders
Brief Title: Platform for the Prospective Mother-child Study of the Determinants of Neurodevelopmental Disorders
Acronym: MARIANNE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Lille (Other); Hospices Civils de Lyon (Other); University Hospital of Saint-Etienne (Other); University Hospital, Rouen (Other); University Hospital, Toulouse (Other); Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0010
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: exposome; child development; genome; risk factors; prenatal cohort
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, hair, nails, baby tooth, stool, blood, umbilical cord blood, placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-Risk Cohort: High family risk cohort for recurrence of autism and other developmental disorders in siblings (have at least one child with a confirmed diagnosis of autism)
  Specific to the High Risk cohort:
  Clinical observations of the unborn child will be performed at 3 months, 6 months, 12 months, between 24 and 30 months, 36 months, and 72 months by psychologists or child psychiatrists in the participating hospitals. They will allow to evaluate the child's behaviors in the areas of communication and social interaction.
  A video recording of the baby at 3 months of age will allow the analysis of the General Movements Assessment.
  If genetic consultation is provided to the family as part of the routine care, the results will be collected and additional blood samples may be taken
  Interventions: Other: Questionnaires; Other: Biospecimen collection; Other: Neurodevelopmental assessment visit; Other: DNA collection
- Low Risk Cohort: Low family risk cohort for recurrence of autism and occurrence of other developmental disorders in siblings. The risk is comparable to the risk observed in the general population (do not have a child with autism, nor with other developmental disorders). Clinical observations of the unborn child will be performed at 72 months by psychologists or child psychiatrists in the participating hospitals, so that children in the "Low family risk" group benefit from the same evaluations as children in the "High family risk" group..
  Interventions: Other: Questionnaires; Other: Biospecimen collection; Other: Neurodevelopmental assessment visit

INTERVENTIONS:
Other: Questionnaires — Parents will be asked to complete online self-questionnaires. These questionnaires will provide essential information on medical data, child development, lifestyle habits, nutritional habits, environmental exposures, and family social characteristics.
Other: Biospecimen collection — urine, hair, nails, baby tooth, stool, blood, umbilical cord blood, placenta
Other: Neurodevelopmental assessment visit — High-Risk Cohort : Clinical observations of the unborn child will be performed at 3 months, 6 months, 12 months, between 24 and 30 months, 36 months, and 72 months by psychologists or child psychiatrists in the participating hospitals. They will allow to evaluate the child's behaviors in the areas of communication and social interaction.
  A video recording of the baby at 3 months of age will allow the analysis of the General Movements Assessment.
  Low-Risk Cohort : linical observations of the unborn child will be performed at 72 months by psychologists or child psychiatrists in the participating hospitals.
Other: DNA collection — If genetic consultation is provided to the family as part of the routine care, the results will be collected and additional blood samples may be taken.
  Groups: High-Risk Cohort

SUMMARY:
Neurodevelopmental disorders such as attention deficit disorder with or without hyperactivity, autism spectrum disorder, language and social communication disorder, motor coordination disorder, learning disorder (dyslexia, dyscalculia, dysorthography), intellectual development disorder are frequent and long-lasting developmental difficulties that can be observed in children in various domains. They are often associated and have a significant impact on daily functioning at school and at home.

The rate of people affected by neurodevelopmental disorders including autism spectrum disorder have increased significantly over the past 20 years. Improved screening only partly explains this evolution.

A genetic predisposition plays an important role in the occurrence of these disorders, however, current scientific data suggest a multifactorial origin. Exposures such as those related to the use of pesticides, air pollution or the presence of endocrine disruptors in our diet could be involved in the genesis of neurodevelopmental disorders, particularly during intrauterine life, a period of great vulnerability.

The current diagnostic pathways for autism rarely enable the early identification of babies at risk. Without early detection and timely targeted intervention, these children have a poor health outcome and do not reach their full potential.

The general objective of the MARIANNE cohort is to constitute a French research infrastructure dedicated to research on the biological and environmental determinants of neurodevelopmental disorders including autism.

This cohort is based on the follow-up of 1200 families with already a child affected by an autism spectrum disorder, which implies a high risk of neurodevelopmental disorders including autism spectrum disorder for the siblings, and of 500 families from the general population with no excess risk of neurodevelopmental disorders. The total number of subjects to be included (mother, father, unborn child and ASD sibling for the HR group) is thus 6300.

The inclusion of these families will be at the beginning of a new pregnancy and the follow-up will be carried out from the second trimester of pregnancy until the children are 6 years old, the age at which the diagnosis of neurodevelopmental disorders is possible.

Biological, clinical, social and environmental data will be collected at different stages of the follow-up and will be included into a large database.

DETAILED DESCRIPTION:
Context: Various forms of Autism Spectrum Disorder (ASD) affect 52 million people worldwide. ASD is an early-onset, life-long and heterogeneous condition believed to arise from combinations of genetic and environmental influences, but without specific known causes. ASD is also a pervasive syndrome that greatly impacts the functioning of the individual throughout life in multiple domains, as well as the family and the broader society. Approximately 1 to 2% of the population is affected by an autism spectrum disorder and 10% to 15% if considering all neurodevelopmental disorders (NDD). They have increased dramatically over the past 20 years, in line with improved screening and diagnostic practices. However, these factors explain only part of the observed increase, and have raised questions about the contribution of environmental changes. Research has shown that ASD overlaps or co-occurs with other clinical neurodevelopmental disorders (NDDs) such as attention-deficit/hyperactivity disorder or intellectual disabilities. This raises the question of phenotypic variations or comorbid association between the disorders. In addition, there is a familial recurrence risk of ASD, studies supporting that younger siblings of children with ASD have an 18 increased relative risk of being diagnosed with ASD themselves. The current diagnostic pathways for ASD rarely enable the early identification of babies at risk. Without early detection and timely targeted intervention, these children have a poor health outcome and do not reach their full potential.

Objectives: The MARIANNE platform is a research infrastructure aiming to allow future scientific studies on the early external (environmental, social) and internal (genetic) drivers of ASD and NDDs, as well as on the outcome of children with ASD.

The primary objective is to compare exposures and development from birth to 6 years of age in children with ASD/NDD and those with normal development in a cohort study whose data will be used to build a large research infrastructure. Specific descriptive, etiological, economic and social objectives are also included:

Descriptive Objectives:

* To identify and clinically characterize cases of ASD and NDD;
* To describe the clinical course of ASD and NDD cases from birth to age 6, in different dimensions (autistic, psychiatric and neurodevelopmental symptoms, health, and development);
* Describe access to care and the care pathway of ASD and NDD cases (use of health services, treatments and interventions) and the modalities of care (specialized interventions, schooling, childcare...).

Etiological Objectives:

* To identify prenatal and perinatal risk factors for ASD and NDD related to the external exposome, such as parental health and lifestyle, socioeconomic characteristics, maternal diet during pregnancy, maternal medication use during pregnancy, pregnancy and delivery complications (clinical, social, health, behaviors, and interventions), and environmental chemical exposures (indoor, outdoor, and occupational);
* To study the interactions between exposome and genome risk factors in ASD or NDD;

Economic and Social Objectives:

* Assess the medico-economic impact of ASD and NDD;
* To study the impact on child health and outcomes of parental mental health, access to care and specialized interventions, socioeconomic status, and education.

Methods:

Cohort study including two groups of families recruited over the same period in the same maternity hospitals, without any other matching criteria.

* At-risk families: 1,200 pregnant women over 18 years of age at increased risk of having a child with TSA or NDDs (e.g. because they already have biological child and/or a partner's biological child with a confirmed ASD), (ii) their partner, and (iii) the future child. The women should be able to read and respond to the questionnaires. Both parents will agree to their child being monitored and to at least the mother being monitored as well.
* Control or Low-risk families: 500 pregnant women, not primiparius (single or multiple pregnancies included from the 2nd trimester of pregnancy), over the age of 18 years, with no biological child over the age of 2 years with a known or suspected diagnosis of ASD or NDD. If there are non-biological children in the family, such as the father's children, the pregnant women may be included in the study if these children have never been suspected of or had a confirmed ASD or NDD. These women should be able to read and respond to the questionnaires. Both parents will agree to their child being monitored and to at least the mother being monitored as well.

The follow-up will start during the second or third trimesters of pregnancy. It will continue at birth and into childhood up until the age of 3 and 6 years, when the diagnoses of ASD and other NDDs can be confirmed by clinical multidisciplinary assessment. Biospecimens (blood, urine…) will be collected from the parents and children and stored in a biobank to allow future assays of exposure and effect biomarkers as well as genotyping. The multidimensional questionnaires and examinations will provide a clinical, biological and social assessment of the child, his/her parents and his/her autistic elder sibling.

Based on the estimated number of subjects needed, 1200 families will be included in the high-risk cohort, which, after a 6-year follow-up, is expected to identify approximately 200 children with ASD, 340 with other ASD, and 660 children with normal development.

The control cohort will consist of 500 families, of which approximately 445 children with normal development, 5 with ASD, and 50 with other NDD are expected. The total number of subjects to be included (mother, father, unborn child and ASD sibling for the HR group) is thus 6300.

Expected benefits: With the recruitment of 1,200 families, MARIANNE cohort is expected to be one of the largest studies on ASD and NDDs with prenatal recruitment. At a societal level, the identification of biomarkers will facilitate the diagnosis and medical management of ASD and NDDs. Another impact covers scientific advances fostered by a better understanding of the underlying etiopathogenic mechanisms. Finally, by proposing an evaluation of the care pathways of a large sample of children, the MARIANNE platform will contribute to providing useful indicators for the piloting of national policies on access to care and management of ASD and NDDs in France.

ELIGIBILITY:
INCLUSION CRITERIA:

General inclusion criteria (High risk and Low risk cohorts)

Mother:

* Be pregnant (single or multiple pregnancy), at least 16 weeks of amenorrhea,
* Have at least one biological child of 24 months or older,
* At least 18 years of age

Father:

* Be the biological father of the unborn child,
* At least 18 years of age

Unborn Child:

- Have a woman study participant as mother.

Specific inclusion criteria for the High risk cohort:

* Autistic sibling: refers to the biological child(ren) of the mother and/or father participating in the study and being the parent(s) of the unborn child
* Be at least 24 months old and less than 18 years old,
* Have a confirmed diagnosis of Autism Spectrum Disorder based on medical records. If in doubt, the SRS-2 (Social Responsiveness Scale for Adults) and PEDS-DM (Parents' Evaluation of developmental status) questionnaires will be completed. Only children with positive scores on one of these questionnaires will be included after validation of the diagnosis by an expert committee,
* In case of several children with Autism Spectrum Disorder based in the siblings, only the last born will be included.

Remarks:

* Autism Spectrum Disorder siblings resulting from a medically assisted procreation are eligible provided that part of the genetic heritage is common to that of the mother or father of the unborn child participating in the study.
* If the father does not live with the mother of the unborn child, his participation is not required and does not preclude the participation of other family members.

EXCLUSION CRITERIA:

General non-inclusion criteria (High risk and Low risk cohorts):

Father and mother:

* Unable to understand French or the study questionnaires
* Participant on protective measures (guardianship or curatorship) or deprived of liberty by judicial or administrative decision, or subject to a legal protection measure
* Not affiliated to a social security system
* Refusal to participate. In the case of consent given for the born and unborn child, the consent must be given by the person(s) with parental authority.
* Live at a distance from the recruitment center incompatible with follow-up.

Specific non-inclusion criteria for the Low risk cohort:

Mother and/or father of unborn child:

- Have a biological child with a diagnosis of Autism Spectrum Disorder or other neuro developmental disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Low risk cohort is a community based sample. High risk cohort is a community based sample as well as an active list of patients followed in specialized department in the management of children with neurodevelopmental disorders.
  The persons involved in the study are the pregnant woman, her partner (if he is the biological father of the unborn child and lives with the mother), the newborn child, and the older sibling with autism.
Sampling Method: Non-Probability Sample
Enrollment: 6300 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2034-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Autism Spectrum Disorder diagnosis | between 60 and 66 months
  ASD diagnosis will be determined by the ADOS-2 (Autism Diagnostic Observation Schedule)
Autism Spectrum Disorder diagnosis | between 24 and 30 months
  ASD diagnosis will be determined by the ADOS-2 (Autism Diagnostic Observation
Developmental Intelligence Disorder diagnosis | at 72 months
  Measure of intelligence quotient by scales adapted to the child's age and level of development and developmental level: Weschler, or Mullen scales
Developmental Coordination Disorder diagnosis | at 72 months
  Description: the diagnosis will be determined by the DCDQ-FE (Developmental Coordination Disorder Parent Questionnaire Coordination), a 15 items scale, which is the French-European version of the DCDQ-0, Developmental Coordination Disorder Parent Questionnaire Coordination to help identify Developmental Coordination Disorder in children aged 5 to 15 years. The items are grouped into three subdomains: 1) control during movement, 2) fine motor/writing, and 3) global coordination. Each item is rated on a 5-point scale, from 1 ("does not match my child at all") to 5 ("matches my child perfectly")."
Attention Deficit Hyperactivity Disorder diagnosis | at 72 months
  The diagnosis will be determined by ADHD-RS, which is a parent questionnaire for the assessment of Attention Deficit Hyperactivity Disorder (ADHD). The items are rated on a 4-point scale (from 0= rarely or never, to 3= very often). A score greater than or equal to 28 is required to qualify as significant ADHD with this scale.
Diagnosis of Language and Learning Disorder | at 72 months
  the diagnosis will be determined with the Parents' Evaluation of developmental status (PEDS: DM), which targets the concerns of parents of children aged 0 to 8 years in 8 domains (gross and fine motor skills and writing and mathematics; social/emotional; oral/written language and reading; adaptive behavior).
  This questionnaire has been validated in several countries and covers several domains, each with 6 to 8 questions and 3 answer choices. The results are evaluated as normal/delayed "Are you worried about your child's development? Yes/No" with details of the reasons, the age of onset and a question on the wish to have an interview with a psychologist or a child psychiatrist.
Socioeconomic and lifestyle risk factors for neurodevelopmental disorders including autism spectrum disorder | at inclusion
  Parental self-questionnaire
Maternal diet and medication use during pregnancy | at inclusion
  Parental self-questionnaire
Environmental exposition | at inclusion
  Parental self-questionnaire. A biological collection is realized for the realization of future assays

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France